CLINICAL TRIAL: NCT07310082
Title: Allograft vs. Autograft to Improve Timely Return to Duty Following Nonunion
Brief Title: Allograft vs. Autograft Nonunion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00140521; HT9425-25-1-0424 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Nonunion Fracture
Keywords: Allograft; Autograft; Nonunion
MeSH Terms: conditions — Fractures, Ununited | interventions — Transplantation, Autologous; Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autograft (Active Comparator): Patients randomized to autograft
  Interventions: Procedure: Autograft
- Allograft (Active Comparator): Patients randomized to allograft.
  Interventions: Procedure: Allograft

INTERVENTIONS:
Procedure: Autograft — Surgeons will decide on the location and method of donor site based on the clinical situation. Most commonly, bone graft will be harvested from the anterior or posterior iliac crest or utilizing the Reamer Irrigator Aspirator in an appropriate long bone. Surgeons may choose to harvest autograft from proximal tibia or distal femur. Donor site location is at the discretion of treating surgeon for patients who randomize to autograft. This treatment arm will not include local autograft only. For large bone defects requiring expansion of autograft with allograft, this will be allowed and recorded. We will use intent-to-treat for statistical analysis of those with allograft expansion of autograft. This autograft will be applied to the nonunion site using the surgeon's typical technique. Internal fixation, revision of fixation, and/or augmentation of fixation will be performed at the discretion of the surgeon.
  Arms: Autograft
Procedure: Allograft — Allograft bone will consist of cancellous or corticocancellous sterile packaged human cadaveric bone. No bone morphogenetic protein, bone marrow aspirate, or other biologic augment will be added. Demineralized bone matrix may be added at the surgeon's discretion. This allograft will be applied to the nonunion site using the surgeon's typical technique. Internal fixation, revision of fixation, and/or augmentation of fixation will be performed at the discretion of the surgeon.
  Arms: Allograft

SUMMARY:
The purpose of this research study is to find out if patients treated for nonunion fracture with autograft or allograft return to activity faster.

DETAILED DESCRIPTION:
The goal of this multi-center prospective randomized controlled trial is to compare short and long-term outcomes of adult patients with long-bone nonunion treated with autograft versus allograft. The main question it aims to answer is: will patients who receive an allograft return to work faster than patients who receive an autograft to treat nonunion fracture.

Participants will be randomized to one of two treatment groups and will complete follow-up surveys during their recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Long bone (tibia, femur, and humerus) nonunion appropriate for either study treatment: to be treated with bone graft harvested from a remote site or using reamer harvester (RIA)
* Nonunion surgery to be performed at least five months after initial fracture fixation
* Prior operative fixation of fracture
* Radiographic apparent bone gap (RABG) of >5cm

Exclusion Criteria:

* Patient that speaks neither English nor Spanish
* Patients whose treatment plan includes local autograft only (available callus from the nonunion site or no planned bone graft)
* Known active infection (defined as any clinical signs or symptoms of active infection, such as fevers, wound redness, warmth, swelling, induration or drainage, and abnormal while blood cell count, erythrocyte sedimentation rate, or C-reactive protein) being treated with antibiotics
* Body mass index greater than 50
* Patients unlikely to follow-up due to homelessness, or planning follow-up at another institution
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic Equivalent for Tasks Score | Week 6
  Time to return to work/duty will be measured using the the International Physical Activity Questionnaire (IPAQ).The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient.
Metabolic Equivalent for Tasks Score | Month 3
  Time to return to work/duty will be measured using the the International Physical Activity Questionnaire (IPAQ).The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient.
Metabolic Equivalent for Tasks Score | Month 6
  Time to return to work/duty will be measured using the the International Physical Activity Questionnaire (IPAQ).The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient.
Metabolic Equivalent for Tasks Score | Month 12
  Time to return to work/duty will be measured using the the International Physical Activity Questionnaire (IPAQ).The IPAQ is a validated, self-report measure that captures detailed information about participation in a wide range of physical activities, including the number of days and amount of time spent in the previous 7 days. Responses for each type of physical activity are then transformed into the number of Metabolic Equivalent for Tasks (METs), and a METs/week is calculated for each patient.
Average Time to Return to Work/Duty | Week 6
  Average number of days it takes for participants to return to work/duty
Average Time to Return to Work/Duty | Month 3
  Average number of days it takes for participants to return to work/duty
Average Time to Return to Work/Duty | Month 6
  Average number of days it takes for participants to return to work/duty
Average Time to Return to Work/Duty | Month 12
  Average number of days it takes for participants to return to work/duty
Number of Participants Returned to Work | Week 6
  Determined by asking whether subjects have returned to work
Number of Participants Returned to Work | Month 3
  Determined by asking whether subjects have returned to work
Number of Participants Returned to Work | Month 6
  Determined by asking whether subjects have returned to work
Number of Participants Returned to Work | Month 12
  Determined by asking whether subjects have returned to work

SECONDARY OUTCOMES:
Percentage of Union | Week 6, Month 3, Month 6, Month 12
  Percentage of union will be assessed via radiographs and determined by the treating surgeon.
Time to Union | Week 6, Month 3, Month 6, Month 12
  Number of days to union
Radiographic Union Scale in Tibial fractures (RUST) score | Month 12
  The RUST score ranges from a minimum score of 4 (definitely not healed) to a maximum score of 12 (completely healed). The final x-ray obtained within a 12-month period following injury will be uploaded to REDCap for review by a blinded panel of investigators from participating sites.
Number of Participants who Return to the Operating Room | Week 6, Month 3, Month 6, Month 12
  Number of participants who return to the Operating Room after procedure
PROMIS-29 Subscale - Physical Function | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means higher physical function.
PROMIS-29 Subscale - Anxiety | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of anxiety.
PROMIS-29 Subscale - Depression | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of depression
PROMIS-29 Subscale - Fatigue | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of fatigue.
PROMIS-29 Subscale - Sleep Disturbance | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of sleep disturbance.
PROMIS-29 Subscale - Pain Interference | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of pain interference.
PROMIS-29 Subscale - Ability to Participate in Social Roles and Activities | Week 6, Month 3, Month 6, Month 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher ability to participate in social roles and activities.
Number of Resource Utilizations | Week 6, Month 3, Month 6, Month 12
  Healthcare utilization, including new hospitalizations, emergency department visits, clinic visits, imaging, and physical therapy sessions will be documented at all follow-up visits
Pain Intensity Scores | Week 6, Month 3, Month 6, Month 12
  Pain will be assessed using the Brief Pain Inventory (BPI). The BPI is a commonly used and validated 15-item measure of pain intensity and interference with daily life. Worst pain score 1-4 = mild pain, 5-6 = moderate pain, 7-10 = severe pain.
Veterans RAND 12 Item Health Survey (VR-12) Scores | Week 6, Month 3, Month 6, Month 12
  The VR-12 is a measure of global health that correspond to seven domains: general health, physical functioning, role limitations, pain, fatigue, social functioning, and mental health. Together, these items are summarized into a Physical Component Score and a Mental Component Score. Scores range from 0-100 with higher scores indicating better physical and mental health functioning.
Work Productivity and Activity Impairment Questionnaire Scores | Week 6, Month 3, Month 6, Month 12
  Participants who report return to work/duty will complete the Work Productivity and Activity Impairment Questionnaire, a validated instrument that measures work time missed and work and activity impairment due to health problems. Measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. The higher number of day equates to more health problems.
Number of Complications | Week 6, Month 3, Month 6, Month 12
  Number of major complications, including infection, implant failure, unplanned or planned return to the operating room related to the nonunion procedure, deep venous thrombosis, or pulmonary embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No